CLINICAL TRIAL: NCT06431529
Title: Exploratory Clinical Study of Tumor Neoantigen-specific T Cells in the Treatment of Advanced Solid Tumors
Brief Title: A Study of Tumor Neoantigen-specific T Cells in the Treatment of Advanced Solid Tumors
Acronym: Neoantigen-T
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: JIANG LONGWEI (Other)
Collaborators: Nanjing University (Other)
Responsible Party: Sponsor-Investigator, JIANG LONGWEI, Associate Researcher, Jinling Hospital, China
Organization: Jinling Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWZL20231008
Record Dates: First submitted 2024-05-22; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Tumor, Solid
Keywords: Solid tumor; T cell; neoantigen
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- tumor neoantigen specific T cell (Experimental): Tumor neoantigen specific T cells will be infused intravenously into patients. The number of T cells will be more than 1.0E9.
  Interventions: Biological: tumor neoantigen specific T cell

INTERVENTIONS:
Biological: tumor neoantigen specific T cell — Isolate the patient's autologous monocytes, induce and culture them into tumor antigen presenting cells in vitro, and then phagocytose tumor tissue cells obtained from biopsy or surgery to present tumor neoantigens to autologous T cells. The final product For tumor neoantigen specific T cells (NeoT).

SUMMARY:
The goal of this clinical trial is to learn if tumor neoantigen-specific T cells can treat patients with advanced solid tumors. The main questions it aims to answer are:

Evaluate the safety of intravenous infusion of tumor neoantigen-specific T cells in the treatment of advanced solid tumors such as ovarian cancer, non-small cell lung cancer, and colorectal cancer.

To evaluate the effectiveness of intravenous infusion of tumor neoantigen-specific T cells in the treatment of advanced solid tumors such as ovarian cancer, non-small cell lung cancer, and colorectal cancer and to study its immunological properties in patients.

DETAILED DESCRIPTION:
In this open, single-armed study, selected patients with advanced solid tumor confirmed by Histopathology will be received tumor neoantigen specific T cells treatment. First, their tumor specimen will be collected from surgery or puncture，then their PBMC will be separated by blood cell separator. This cells will be cultured and selected in GMP laboratory to make tumor neoantigen specific T cells. The tumor neoantigen specific T cells will be infused intravenous into patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Patients with solid malignant tumors confirmed by histology or cytology such as ovarian cancer, non-small cell lung cancer or colorectal cancer;
3. Cancer patients who have failed previous standard treatments or who have refused subsequent chemotherapy and whose expected survival time exceeds 3 months;
4. ECOG: 0-2 points;
5. Patients of childbearing age need to take appropriate protective measures (contraceptive measures or other birth control methods) before enrollment and during the experiment;
6. Those who can understand this trial and have signed the informed consent form;
7. Able to follow the research protocol and follow-up procedures

Exclusion Criteria:

1. Those who have received any form of immunotherapy within the past 3 months;
2. Those who need to use immunosuppressants;
3. Those who have received anti-tumor treatment such as tumor chemotherapy, radiotherapy, and secondary and above surgery within the past month;
4. Those who have a history of other tumors in the past, unless it is cervical cancer in situ, treated squamous cell carcinoma or bladder epithelial tumor (Ta and TIS), or other malignant tumors that have received radical treatment (at least 5 years before enrollment) );
5. White blood cell count <3E9/L, platelet count <80E9/L;
6. AST and ALT>3×the upper limit of normal (ULN), total bilirubin>2×ULN, and AST and ALT>6×ULN in patients with liver metastasis;
7. Creatinine clearance <60ml/min;
8. Abnormal coagulation function;
9. The patient has active bacterial or fungal infection (≥Grade 2 of NCI-CTC, third edition);
10. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive and the peripheral blood hepatitis B virus (HBV) DNA detection value is >100 IU/mL; hepatitis C virus (HCV) antibody is positive and the peripheral blood hepatitis C Those who are positive for hepatitis virus (HCV) RNA; those who are positive for human immunodeficiency virus (HIV) antibodies; those who are positive for cytomegalovirus (CMV) DNA; those who are positive for syphilis;
11. Diseases judged by the researcher to be ineligible for inclusion: including but not limited to severe liver, kidney or metabolic diseases requiring drug treatment, uncontrollable coronary artery disease or asthma, and uncontrollable cerebrovascular disease.
12. Women who are pregnant or breastfeeding, and women of childbearing age must have a negative pregnancy test within 7 days before enrollment;
13. Substance abuse, clinical or psychological or social factors that affect informed consent or research implementation;
14. Those who may be allergic to study drugs;
15. Participate in other clinical trials one month before registration;
16. Patients who cannot undergo mononuclear cell separation or whose peripheral venous access cannot be opened;
17. Any uncertain factors that affect patient safety or compliance;
18. Other researchers believe that the subject is not suitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety of tumor neoantigen specific T cells in the treatment of advanced tumor patients | 2 years
  The adverse events and severe adverse events will be evaluated.

SECONDARY OUTCOMES:
Evaluate the efficiency of tumor neoantigen specific T cells in the treatment of advanced solid tumor. | 2 years
  The objective clinical response will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shaochang, MD, Study Director — Jinling Hospital, China
Locations (1):
- Nanjing Jinling Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No